CLINICAL TRIAL: NCT03490890
Title: Microwave Ablation in Ground Glass Nodules
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xin Ye, Principal Investigator, Shandong Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shandong PH JN
Record Dates: First submitted 2018-03-26; First posted 2018-04-06 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Microwave Ablation; Lung Cancer
Keywords: microwave ablation; lung cancer; ground glass nodules
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: All patient with GGO were treated with microwave ablation
Masking Description: All patient with GGO were treated with microwave ablation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microwave ablation in the GGO (Experimental): Patients with GGO were treated with microwave ablation.
  Interventions: Other: Microwave ablaton

INTERVENTIONS:
Other: Microwave ablaton — Patients with pathology verified GGO were treated with MWA.

SUMMARY:
GGO was commonly observed recently.Radiofrequency ablation has been widely applied in the treatment of patients with GGO. No study had explored the microwave ablation in the treatment of GGO.

DETAILED DESCRIPTION:
GGO was common with the development of image. Treatments of GGO include radical surgery and irradiation. For patients who were poor candidate of surgery, image guided thermal ablation could be an alternative.Radiofrequency ablation has been widely applied in the treatment of eary-stage non small cell lung cancer and those patients with GGO. However, up to date, no study had explored the microwave ablation in the treatment of GGO.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a histologically verified AIS or MIA.
2. The tumors small enough to treat (usually ≤3 cm), and without chest pleura invasion.
3. Solid cements in the GGO less than 50%.
4. No other sites of disease observed.
5. Patient is not a candidate for surgical removal of the cancer, or refused surgery.
6. Patient is not a candidate for radiation therapy, or refused radiation therapy.
7. Patient has > 6 month life expectancy.
8. Eastern Cooperative Oncology Group performance status of 0 to 2.
9. No prior anticancer treatments including surgery, radiation,chemotherapy or local treatments.
10. Sufficient organ functions.
11. Written informed consent.

Exclusion Criteria:

1. Active bacterial or fungous infection.
2. Simultaneous or metachronous (within the past 5 years) double cancers.
3. Women during pregnancy or breast-feeding.
4. Interstitial pneumonitis, pulmonary fibrosis, or severe pulmonary emphysema.
5. Uncontrollable diabetes mellitus. History of severe heart disease, heart failure, myocardial infarction within the past 6 months or attack of angina pectoris within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
The survival of patients with GGO treated with MWA | From the date of randomization until the date of the date of death from any cause, assessed up to 60 months
  The overall survival

SECONDARY OUTCOMES:
The disease free survival of patients with GGO treated with MWA | From date of randomization until the date of first documented progression, assessed up to 60 months
  The disease free survival

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year
  The safety

CONTACTS AND LOCATIONS:
Overall Officials: Xin Ye, Study Director — Shandong Provincial Hospital
Locations (15):
- China (15):
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Dezhou People's Hospital, Dezhou, Shandong
  - The Second People's Hospital of Dezhou, Dezhou, Shandong
  - Jinan Military General Hospital, Jinan, Shandong
  - Affliated Hospital of Shandong Academy of Medical Sciences, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Provincial Hospital affliated to Shandong University, Jinan, Shandong
  - Affliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng Cancer Hospital, Liaocheng, Shandong
  - The People's Hospital of Pingyi Country, Linyi, Shandong
  - Affliated Hospital of Taishan Medical University, Taian, Shandong
  - The People's Liberation Army 88 Hospital, Taian, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Tengzhou center of people's hospital, Zaozhuang, Shandong

IPD SHARING:
Plan to Share IPD: No